CLINICAL TRIAL: NCT01042496
Title: 1H-MR Spectroscopy of Bipolar Depression Before and After Lamotrigine Treatment
Brief Title: Bipolar Depression Before and After Lamotrigine Treatment
Acronym: 1HMRS-BP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark Frye, M.D., Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-004163; R01MH079261-01A2 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Bipolar Depression
Keywords: Bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bipolar Group (Active Comparator): Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC) before and after treatment with Lamotrigine.
  Interventions: Drug: Lamotrigine; Procedure: 1H-MR
- Control Group (Active Comparator): Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC).
  Interventions: Procedure: 1H-MR

INTERVENTIONS:
Drug: Lamotrigine — 12 week open trial: 25mg/day for 2 weeks, 50mg/day for 2 weeks, 100mg/day for 2 weeks, 200mg/day for 6 weeks. Flexible titration for early response and/or side effects.
  Other Names: Lamictal®
  Arms: Bipolar Group
Procedure: 1H-MR — Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC).

SUMMARY:
This study compared glutamate and other neurometabolites measured by proton magnetic resonance spectroscopy (1H-MRS) in bipolar I and II patients currently depressed with age-matched healthy controls. The study will also compare 1H-MRS of bipolar I and II patients before and after taking a 12-week course of lamotrigine.

The goal of this study was to better understand the neurobiology of bipolar depression and how lamotrigine may therapeutically impact brain function and mood response.

The hypothesis was that in comparison to non-remission participants, bipolar participants who achieve remission (defined as a Montgomery Asberg Depression Rating Scale (MADRS) score <12 at week 12) associated with lamotrigine monotherapy will exhibit a greater decrease in glutamate (Glu) and an increase in N-acetyl aspartate (NAA), reported as a cerebrospinal fluid (CSF)-corrected absolute concentration percent change from baseline to endpoint in anterior cingulate (AC) and dorsolateral prefrontal cortex (DLPFC).

DETAILED DESCRIPTION:
Depression is the predominant prevailing mood state in bipolar disorder and bipolar depression is associated with substantial morbidity and mortality. However, in comparison to acute mania, bipolar depression is understudied both from the standpoint of its pathophysiology as well as clinical trials which include FDA-approved treatments. Given this lack of evidence to base guidelines, clinicians and patients are limited as to how best to treat the depressive phase of the illness.

Proton magnetic resonance spectroscopy (1H-MRS) is a valuable, non-invasive method to study in-vivo brain biochemistry. Of the novel imaging paradigms, MRS is uniquely positioned to investigate biochemical mechanism of drug action that is objectively measurable and clinically relevant. As there is increasing interest in glutamatergic dysregulation in mood disorders, this project will utilize 1H-MRS to study glutamate and glutamine levels in brain regions implicated in bipolar disorder (anterior cingulate and dorsolateral prefrontal cortex).

This was a 5-year single-site study of bipolar depression utilizing 1H-MR spectroscopy before and after treatment with lamotrigine. At baseline bipolar depressed subjects and age-matched controls underwent a 1H-MRS at Mayo Clinic in Rochester, Minnesota. The bipolar depressed subjects were then be placed on 12-week, open evaluation of lamotrigine monotherapy. After 12 weeks, the bipolar subjects underwent a second 1H-MRS scan.

Two different MRS sequences were used to measure the brain chemicals in a single 2 x 2 x 2 cm cube located in the center of anterior cingulate cortex: an intermediate echo-time PRESS sequence and a 2D J-resolved averaged PRESS sequence. Spectroscopic data were inspected for quality; subjects whose data were contaminated by artifact were excluded from the study. Spectra were then processed using LCModel to quantify brain chemical levels. Regular brain MRI images were segmented, yielding a map of the amount of CSF in the head. The MRS cube was overlaid onto the CSF map and the fraction of CSF within the cube measured. This measurement was used to "remove" the CSF from the MRS cube giving brain chemical concentrations. The concentrations were then used for statistical analysis.

Note: All of the spectroscopy data are expressed in Institutional Units (IU).

ELIGIBILITY:
Bipolar Group Inclusion Criteria:

* Diagnosis of Bipolar Type I or II disorder depress phase (SCID confirmed)
* Moderate depression as confirmed by Montgomery Asberg Depression Rating Scale greater than or equal to 20
* Negative urine toxicology screen
* Negative urine pregnancy test
* No clinically significant lab abnormalities for complete blood count (CBC), Thyroid stimulating hormone (TSH), Sodium (Na+), Potassium (K+), Chlorine (Cl-), Carbon dioxide (CO2), creatinine (CREA), blood urea nitrogen (BUN), Glucose, hepatic panel.

Bipolar Group Exclusion Criteria:

* Inability to provide informed consent
* Any current Axis I diagnosis other than anxiety disorders needing concurrent antidepressant therapy
* History of active substance abuse/dependence within the last 3 months
* History of claustrophobia
* History of adverse reaction to Lamotrigine
* Fluoxetine and decanoate antipsychotic therapy
* Unwilling or unable to taper current sub-optimal psychotropic medications other than a stable dosage of Lithium, Depakote, or an Atypical Antipsychotic approved by study personnel
* Unstable active medical illness
* Pregnancy or breast-feeding
* Male/ Female not practicing a reliable form of birth control (condom, Intrauterine Device (IUD), depo injection)
* Female wishing to commence oral contraceptive therapy within 3 months of enrollment date (stable oral contraceptive therapy exception)
* Active suicidal ideation with plan
* History of major head trauma with loss of consciousness > 5 minutes or skull fracture
* History of previous neurological event (epilepsy, stroke, transient ischemic attack)
* Implanted metal objects (i.e., pacemakers, aneurysm clips, metal prostheses, joints, rods)
* Inability to speak English
* Prominent Axis II disorder [This will be assessed by the principal investigator, who has >10 years clinical experience with this population. Hospital discharge summaries and outpatient medical records will be reviewed for evidence that Axis II pathology is the primary psychiatric disturbance (i.e., adequate trials of mood stabilizing treatments with minimal to no response, prominent self injurious behavior in the absence of significant mood symptomatology, or atypical cycle patterns)].

Healthy Control Group Inclusion Criteria:

* Negative urine toxicology screen
* Negative urine pregnancy test
* Normal blood values for thyroid stimulating hormone (TSH)

Healthy Control Group Exclusion Criteria:

* Inability to provide informed consent
* Any current Axis I or II diagnosis
* Known history of claustrophobia
* Lifetime personal or family history (first-degree relative) of dementia, substance-related disorder (nicotine abuse or dependence exception), psychotic disorder, mood disorder (history of bereavement exception), anxiety disorder (specific phobia exception)
* Unstable active medical illness
* Pregnancy or breast-feeding
* Male /Female not practicing a reliable form of birth control (condom, IUD, depo injection)
* History of major head trauma with loss of consciousness > 5 minutes or skull fracture
* History of previous neurological event (epilepsy, stroke, transient ischemic attack)
* Implanted metal objects (i.e., pacemakers, aneurysm clips, metal prostheses, joints)
* Inability to speak English
* On current medications known to affect glutamate (i.e., Riluzole).
* Any medically remarkable impairment due to a medical condition or brain injury resulting in significant impairment in cognitive functioning based on neuropsychological test battery and/or MRS scan results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: 39 subjects signed informed consent for the Bipolar Group, but 9 were screen failures, and one subject signed consent but did not start the study. 33 subjects signed informed consent for the Healthy Control group, and all of these subjects completed the study.
Period: Overall Study
Arm/Group | Bipolar Group | Control Group
Started | 29 | 33
Completed | 29 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who took part in the study were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bipolar Group | Control Group | Total
Number analyzed (Participants) | 29 | 33 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.10 (13.44) | 35.18 (10.1) | 35.61 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 12 | 18 | 30
Region of Enrollment [Number; unit: participants]
  United States | 29 | 33 | 62

OUTCOME MEASURES:

1. Primary Outcome: Mean Montgomery-Åsberg Depression Rating Scale (MADRS) Score at Baseline for Both Groups, and After 12 Weeks of Lamotrigine Monotherapy for the Bipolar Group
Description: The MADRS is a 10-item observer rating scale assessing symptoms of depression. The score ranges from 0 (no depression) to 60 (very depressed). A score of less than 12 is considered clinical remission of depression.
Time Frame: baseline, 12 weeks
Population: The control group only did the MADRS depression rating scale at baseline. 25 participants in the Bipolar group took the MADRS depression rating scale at 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bipolar Group | Control Group
Number analyzed (Participants) | 29 | 33
units on a scale
  Baseline | 27.79 (5.80) | 0.30 (0.64)
  12 weeks | 14.28 (11.67) | NA (NA) — The control group only did the MADRS depression rating scale at baseline.

2. Secondary Outcome: Glutamate+Glutamine (GLX) Measured in Mid Anterior Cingulate Cortex (MACC) & Left Dorsal Lateral Prefrontal Cortex (LDLPC) Using Long TE PRESS MRS Technique at Baseline for Both Groups; After 12 Weeks of Lamotrigine Monotherapy for the Bipolar Group
Description: Two different MRS sequences were used to measure the brain chemicals in in anterior cingulate and left dorsal lateral prefrontal cortex : an intermediate echo-time PRESS sequence and a 2D J-resolved averaged PRESS sequence. (Note: The intermediate echo-time PRESS sequence was used for this outcome measure.) Spectroscopic data were inspected for quality; subjects whose data were contaminated by artifact were excluded from the study. Spectra were then processed using LCModel to quantify brain chemical levels. Regular brain MRI images were segmented, yielding a map of the amount of cerebrospinal fluid (CSF); the MRS voxel was overlaid onto the CSF map and the fraction of CSF was measured. This CSF corrected measurement was used for statistical analysis.
Time Frame: baseline, after 12 weeks
Population: Sample sizes varied due to imaging results/scan viability. Excessive noise resulted in poor metabolite readings which in-turn were not used in the final analysis. Baseline: control group MACC n=7, LDLPC n=8, Bipolar group MACC n=18, LDLPC n=27. Bipolar group 12 weeks MACC n=12, LDLPC n=16. The control group did not do the procedure at 12 weeks.
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Arm/Group | Bipolar Group | Control Group
Number analyzed (Participants) | 28 | 8
Institutional Units (IU)
  Baseline GLX measured in MACC | 15.08 (3.88) | 11.98 (2.06)
  12 Weeks GLX measured in MACC | 12.69 (4.05) | NA (NA) — The control group did not do the procedure at 12 weeks.
  Baseline GLX measured in LDLPC | 14.0 (2.7) | 12.9 (1.4)
  12 Weeks GLX measured in LDLPC | 14.1 (2.7) | NA (NA) — The control group did not do the procedure at 12 weeks.

3. Secondary Outcome: N-acetylaspartic Acid (NAA) Measured in the MACC and LDLPC Using the Long TE (TE80) PRESS MRS Technique at Baseline for Both Groups, and After 12 Weeks of Lamotrigine Monotherapy for the Bipolar (BP) Group and BP Responders and Non-responders
Description: Two different MRS sequences were used to measure the brain chemicals in a single 2 x 2 x 2 cm cube located in the center of anterior cingulate cortex: an intermediate echo-time PRESS sequence and a 2D J-resolved averaged PRESS sequence. (Note: The intermediate echo-time PRESS sequence was used for this outcome measure.) Spectroscopic data were inspected for quality; subjects whose data were contaminated by artifact were excluded from the study. Spectra were then processed using LCModel to quantify brain chemical levels. Regular brain MRI images were segmented, yielding a map of the amount of CSF in the head. The MRS voxel was overlaid onto the CSF map and the fraction of CSF within the voxel measured. This CSF-corrected measurement was used for statistical analysis.
Time Frame: baseline, 12 weeks
Population: Samples varied due to imaging results/scan viability. Baseline: control group MACC (M) and LDLPC (L) n=8, BP whole M n=28 (3 didn't complete), L n=27, BP Responders M n=13, L n=11, BP nonresponders M and L n=12; BP whole 12 weeks M and L n=16. BP Responders M and L n=10, BP nonresponders M and L n=6. Controls didn't do the procedure at 12 weeks.
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Groups:
- Bipolar Lamotrigine Responders Group: Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC) before and after treatment with Lamotrigine.
  Lamotrigine: 12 week open trial: 25mg/day for 2 weeks, 50mg/day for 2 weeks, 100mg/day for 2 weeks, 200mg/day for 6 weeks.
  1H-MR: Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC).
- Bipolar Lamotrigine Non-Responders Group: Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC) before and after treatment with Lamotrigine.
  Lamotrigine: 12 week open trial: 25mg/day for 2 weeks, 50mg/day for 2 weeks, 100mg/day for 2 weeks, 200mg/day for 6 weeks. Flexible titration for early response and/or side effects.
  1H-MR: Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC).
  Non-responders were those bipolar participants who did not achieve remission (defined as a Montgomery Asberg Depression Rating Scale (MADRS) score <12 at week 12).
- Bipolar Lamotrigine Group as Whole: Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (DLPFC) before and after treatment with Lamotrigine.
  Lamotrigine: 12 week open trial: 25mg/day for 2 weeks, 50mg/day for 2 weeks, 100mg/day for 2 weeks, 200mg/day for 6 weeks.
  1H-MR: Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (DLPFC).
Arm/Group | Bipolar Lamotrigine Responders Group | Control Group | Bipolar Lamotrigine Non-Responders Group | Bipolar Lamotrigine Group as Whole
Number analyzed (Participants) | 13 | 8 | 12 | 28
Institutional Units (IU)
  LDLPC Baseline NAA | 19.5 (1.9) | 20.1 (1.5) | 21.0 (2.8) | 20.0 (2.5)
  LDLPC 12 weeks NAA | 20.3 (2.1) | NA (NA) — The control group did not do the procedure at 12 weeks. | 20.8 (2.9) | 20.5 (2.4)
  MACC Baseline NAA | 15.7 (2.9) | 17.51 (1.77) | 15.2 (3.3) | 15.4 (3.0)
  MACC 12 weeks NAA | 14.3 (3.2) | NA (NA) — The control group did not do the procedure at 12 weeks. | 14.9 (3.8) | 14.5 (3.4)

4. Secondary Outcome: Mean Glutamate (GLU) Measured in the MACC and LDLPC Using the ProFit MRS Technique at Baseline for Both Groups, After 12 Weeks of Lamotrigine Monotherapy for the Bipolar Group
Description: Two different MRS sequences were used to measure the brain chemicals in a single 2 x 2 x 2 cm cube located in the center of anterior cingulate cortex: an intermediate echo-time PRESS sequence and a 2D J-resolved averaged PRESS sequence. (Note: The 2D J-resolved averaged PRESS sequence was used for this outcome measure.) Spectroscopic data were inspected for quality; subjects whose data were contaminated by artifact were excluded from the study. Spectra were then processed using LCModel to quantify brain chemical levels. Regular brain MRI images were segmented, yielding a map of the amount of CSF in the head. The MRS voxel was overlaid onto the CSF map and the fraction of CSF within the voxel measured. This CSF-corrected measurement was then used for statistical analysis.
Time Frame: baseline, 12 weeks
Population: Sample sizes varied due to imaging results/scan viability. Excessive noise resulted in poor metabolite readings which in-turn were not used in the final analysis. Baseline: control group MACC n=8, LDLPC n=8, Bipolar group MACC n=13, LDLPC n=13. Bipolar group 12 weeks MACC n=8, LDLPC n=17. The control group did not do the procedure at 12 weeks.
Measure: Mean (Standard Deviation); unit: Institutional Units (IU)
Groups:
- Control Group: Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (DLPFC).
  1H-MR: Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (DLPFC).
Arm/Group | Bipolar Group | Control Group
Number analyzed (Participants) | 17 | 8
Institutional Units (IU)
  Baseline MACC | 147.55 (32.57) | 157.51 (36.17)
  12 Weeks MACC | 134 (13.5) | NA (NA) — The control group did not do the procedure at 12 weeks.
  Baseline LDLPC | 65.4 (15.5) | 64.1 (12.6)
  12 Weeks LDLPC | 63.5 (11.6) | NA (NA) — The control group did not do the procedure at 12 weeks.

5. Secondary Outcome: Glutamine/Glutamate Ratio Measured in the LDLPC at Baseline Using the ProFit Magnetic Resonance Spectroscopy (MRS) Technique
Description: as for outcome 4
Time Frame: baseline
Population: Sample sizes varied between both scanning locations LDLPC and MACC and between metabolites due to imaging results/scan viability. Some subject scans yielded more viable information/ less noise during the scan process. Excessive noise resulted in poor metabolite readings which in-turn were not used in the final analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bipolar Group | Control Group
Number analyzed (Participants) | 6 | 0
ratio | 1.27 (.62) |

ADVERSE EVENTS:
Groups:
- Bipolar Group: Subjects underwent proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC) before and after treatment with Lamotrigine.
  Lamotrigine: 12 week open trial: 25mg/day for 2 weeks, 50mg/day for 2 weeks, 100mg/day for 2 weeks, 200mg/day for 6 weeks
  1H-MR: Proton magnetic resonance spectroscopy (1H-MR) evaluation of medial anterior cingulate cortex (MACC) and left dorsal lateral prefrontal cortex (LDLPC).
Arm/Group | Bipolar Group | Control Group
Serious Adverse Events (participants affected / at risk) | 5/29 | 0/33
Other Adverse Events (participants affected / at risk) | 6/29 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Group (N=29) | Control Group (N=33)
Hospitalization due to progression of disease (Psychiatric disorders) | 1 (1) | 0 (0)
Admitted to ER due to symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Death (Psychiatric disorders) | 1 (1) | 0 (0)
Worsening of bipolar symptoms (Psychiatric disorders) | 1 (1) | 0 (0)
Withdrawal from study due to decrease in mood (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Group (N=29) | Control Group (N=33)
Bruise on back of head near ossiput (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swollen lymph node (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rash on left knee (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abnormal high AST level at study exit (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abnormal high GGT level at study exit (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Paresthesia of Right Shoulder Blade (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes